CLINICAL TRIAL: NCT07078032
Title: A Randomized Controlled Trial Evaluating the Effectiveness of a Novel Risk-Stratified Screening Strategy for Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20250711
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prediction Model Arm (Experimental): Lung Cancer Risk Prediction Model Arm
  Interventions: Diagnostic Test: Prediction Model Arm
- Standard Screening Arm (Active Comparator): Traditional High-Risk Factors Arm
  Interventions: Diagnostic Test: Standard Screening Arm

INTERVENTIONS:
Diagnostic Test: Prediction Model Arm — Lung cancer risk stratification via prediction model integrating: advanced age, lung cancer family history, personal cancer history, childhood coal exposure, asthma history, and food allergy history. High-risk individuals receive LDCT screening. Thoracic physicians guide management of screen-positive cases.
  Other Names: Lung Cancer Risk Prediction Model Arm
  Arms: Prediction Model Arm
Diagnostic Test: Standard Screening Arm — Participants are screened based on NCCN guideline criteria. High-risk individuals receive LDCT screening. Thoracic physicians guide management of screen-positive cases.
  Other Names: Traditional High-Risk Factors Arm
  Arms: Standard Screening Arm

SUMMARY:
A nationwide population-based multi-center RCT enrolling ≥60,000 eligible residents to compare screening effectiveness between risk-prediction-model-driven and traditional guideline-based high-risk lung cancer screening strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Residents with local household registration residing continuously in the region for ≥3 years.
2. Aged 40-74 years at enrollment.

Exclusion Criteria:

1. Prior diagnosis of lung cancer (histologically/cytologically confirmed)
2. Currently receiving active treatment for any malignancy.
3. Presence of severe comorbidities with life expectancy <5 years
4. Participation in any lung cancer screening program within 5 years.
5. Functional dependency (ADL score ≤2) OR unwillingness to comply with protocol-required follow-up.
6. Declined to provide written informed consent.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) of Screening Strategies | From enrollment through completion of diagnostic confirmation (up to 3 months post-screening)
  Proportion of true lung cancer cases among participants with positive screening results, confirmed by histopathology within 3 months after screening. Calculated as: (True Positives) / (True Positives + False Positives) × 100%. Assessed separately for both screening arms.

SECONDARY OUTCOMES:
Sensitivity of Screening Strategies | From screening to 12-month follow-up
  Proportion of true lung cancer cases correctly identified by screening, confirmed through histopathology within 6 months. Calculated as: True Positives / (True Positives + False Negatives) × 100%. Includes interval cancers detected within 12 months post-screening
Specificity of Screening Strategies | From screening to 12-month follow-up
  Proportion of cancer-free participants correctly identified as screening-negative. Calculated as: True Negatives / (True Negatives + False Positives) × 100%. Cancer-free status confirmed by 12-month follow-up
Negative Predictive Value (NPV) | From screening to 12-month follow-up
  Proportion of screening-negative participants without lung cancer. Calculated as: True Negatives / (True Negatives + False Negatives) × 100%. Absence of cancer confirmed by 12-month follow-up including LDCT and clinical evaluation.
Early-Stage Shift Proportion | At time of cancer diagnosis (within 3 months post-positive screening)
  Percentage of screen-detected lung cancer cases diagnosed at early stage (AJCC 8th ed. Stage I-II) versus late stage (Stage III-IV). Calculated as: (Early-stage cases) / (Total screen-detected cases) × 100%.
Lung Cancer-Specific Mortality Rate | From randomization to 3-year follow-up
  Death rate attributable to lung cancer, verified by independent mortality review committee using ICD-10 codes (C34.0-C34.9) and medical records. Expressed as deaths per 1,000 person-years.
Overall Survival in Screen-Detected Lung Cancer | From cancer diagnosis to 3-year follow-up
  Time from pathological diagnosis of lung cancer to death from any cause. Assessed using Kaplan-Meier method with censoring at last follow-up. Reported as median survival with 95% CI.

IPD SHARING:
Plan to Share IPD: No